CLINICAL TRIAL: NCT03708068
Title: Early Exclusive Enteral Nutrition in Stable Preterm Infants at 30 0/7 - 33 6/7 Weeks Gestation: A Randomized Controlled Trial
Brief Title: Early Exclusive Enteral Nutrition in Early Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belal Alshaikh (Other)
Responsible Party: Sponsor-Investigator, Belal Alshaikh, Neonatologist, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB18-0772
Record Dates: First submitted 2018-10-01; First posted 2018-10-16 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Enteral Nutrition
Keywords: Exclusive; Enteral Nutrition; Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Exclusive Enteral Nutrition (Experimental): Feeds will start at least at 80% of reference daily fluid intake from day one of life.
  Feeds will be advanced by 20-30 ml/kg per day on second day onwards until infant reaches full enteral feed.
  Interventions: Other: Early exclusive enteral nutrition
- Conventional Enteral Nutrition (No Intervention): Infants will be fed as per current Neonatal Intensive Care Unit feeding tables:
  1. Infants with birth weight 1000-1500 g will be fed on 15-20 ml/kg human milk in day one. Feeds will be advanced by 15-20 ml/kg per day on second day onwards until infant reaches full enteral feeds.
  2. Infants with birth weight >1500 g will be started on 20-30 ml/kg per day on day one. Feeds will be advanced by 20-30 ml/kg per day on second day onwards until infant reaches full enteral feeds.

INTERVENTIONS:
Other: Early exclusive enteral nutrition — Infants will be fed at least 80% of reference daily fluid intake from day one. Feeds will be advanced by 20-30 ml/kg per day on second day onwards to meet reference daily fluid intake until infant reaches full enteral feed.
  Other Names: Early Total Enteral Feed
  Arms: Early Exclusive Enteral Nutrition

SUMMARY:
Enteral nutrition in preterm infants is usually started and advanced slowly until reaching full enteral feeds. Most preterm infants born before 34 weeks gestation require parenteral fluids to maintain normal blood sugar level and prevent excessive weight loss and dehydration. Availability of donor human milk (DHM) along with low incidence of necrotizing enterocolitis (NEC) in preterm infants born at 30-33 weeks have encouraged neonatologists to start feeding early and advance it faster in order to shorten time on parenteral nutrition (PN) and minimize the need for intravenous access. The objectives of this trial is to study whether exclusive enteral nutrition from day of birth (i.e. no PN) results in shorter time to achieve full enteral feed when compared with traditional feeding regimen that involves a combination of PN and progressive enteral feeding.

DETAILED DESCRIPTION:
Early nutritional support of preterm infants born at 30-33 weeks gestation is usually achieved via a combination of parenteral nutrition (PN) and enteral feeding that is advanced over few days to reach full enteral feed. Recent studies suggest that rapid increase of enteral feed volumes results in shorter duration on PN and earlier achievement of full enteral feed without increasing the risk of necrotizing enterocolitis (NEC) or death. Although PN has an important role in nutrition of preterm infants, it is associated with increased risk of metabolic and infectious complications even when it is used for a short period of time. Furthermore, PN mandates the need for peripheral or central intravenous access. Provision of full enteral feed volume that meets reference daily fluid intake from day of birth is used frequently and successfully in stable preterm infants born after 33 weeks. Expanding the use of this regimen to stable preterm infants born at 30-33 weeks gestation may help avoid unnecessary start of intravenous access, prevent complications related to PN, and encourage mother-infant bonding experience.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born at 30 0/7 - 33 6/7 weeks gestation
2. Birth weight greater than 1000 g
3. Consent to use donor human milk
4. Postnatal age is less than 48 hours from birth
5. Infant is ready to start on feeding (as per clinical team) or feeding volume, when already started, is ≤12 ml/kg per day (total) and/or the infant received ≤2 feeds based on current feeding policy or physician descrition (total volume of the received feeds is ≤20 ml/kg per day).

Exclusion Criteria:

1. Cord PH < 7.00 or Cord base access (BE) < -16
2. Apgar score < 7 at 5 minute
3. Lactate level ≥3 (if done for clinical indication)
4. Need for positive pressure ventilation (PPV) for >1 minute.
5. Hemodynamic instability (hypotension or poor perfusion at any time in this 48 hours)
6. Small for gestational age <3 percentile on Fenton chart and/or fetal absent or reversed umbilical arterial end-diastolic blood flow.
7. Major congenital malformation
8. Symptomatic or severe hypoglycemia (blood glucose <1.8 mmol/L)
9. Infants with moderate to severe respiratory distress.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Duration to achieve of full enteral feeds in days | Till 30 days of life
  Day of life to achieve full enteral feeding defined as 140 ml/kg/day which is sustained for at least 3 days

SECONDARY OUTCOMES:
Length of hospital stay | At discharge from neonatal intensive care unit (NICU), up to 90 days of life
  Length of hospital stay in days
Feeding intolerance | Till 30 days of life
  Presence of one or more of the following:
  1. vomiting more than 2 times during any 24 h period,
  2. any episode of bile- or blood-stained vomiting,
  3. abdominal wall erythema or tenderness that resulted in cessation of feed.
Incidence of late onset sepsis | At discharge from NICU, up to 90 days of life
  Any microbial growth in blood, cerebrospinal fluid or urine after 72 hours of admission in NICU
Incidence of NEC | At discharge from NICU, up to 90 days of life
  Any Stage II and above according to Bell's staging criteria
Incidence of hypoglycemia | Till 30 days of life
  Defined as point of care testing Glucose < 2.6 mmol/L at any time after rollment in study

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Peter Lougheed Hospital, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta

REFERENCES:
- [Derived] Alshaikh BN, Hassan O, Alburaki W, Dharel D, Elsharkawy A, Singal N, Yusuf K, Awad EA. Early exclusive enteral feeding in 30-33 weeks gestation infants: a randomized controlled trial. J Perinatol. 2025 May;45(5):628-634. doi: 10.1038/s41372-025-02217-0. Epub 2025 Feb 2. PMID 39894877